CLINICAL TRIAL: NCT02067013
Title: Analysis of Vitreous and Aqueous Humor for Ocular Growth Factors, Cytokines, Chemokines, and Ranibizumab Pharmacokinetics Associated With Various Retinal Disease
Brief Title: Analysis of Aqueous and Vitreous Humor
Acronym: ARK
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: California Retina Consultants (Other)
Responsible Party: Principal Investigator, Robert Avery, Principal Investigator, California Retina Consultants
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ML28894s
Record Dates: First submitted 2014-02-17; First posted 2014-02-20 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Proliferative Diabetic Retinopathy; Macular Degeneration; Macular Hole; Neovascular Glaucoma
Keywords: Tractional retinal detachment; Exudative retinal detachment; Macular hole; Neovascular glaucoma
MeSH Terms: conditions — Macular Degeneration; Retinal Perforations; Glaucoma, Neovascular | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab (Active Comparator): Subjects undergoing surgery for neovascular glaucoma, diabetic retinopathy, or tractional Retinal Detachment due to AMD will receive one intravitreal injection of ranibizumab within 2 weeks of their surgery. Vitreous and aqueous humor samples will be collected during the surgery. Serum samples may be collected before, during, or after surgery.
  Interventions: Drug: Ranibizumab
- Control (Placebo Comparator): Subjects undergoing surgery for ERM or macular hole will NOT receive an injection of ranibizumab, but will have vitreous, and aqueous humor samples collected during surgery (no serum collection).
  Interventions: Other: No Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Subjects in the Ranibizumab arm will receive an injection of drug within 2 weeks prior to their surgery.
  Other Names: Lucentis
  Arms: Ranibizumab
Other: No Ranibizumab — Subjects in the control arm will NOT receive an injection of drug within 2 weeks prior to their surgery.
  Arms: Control

SUMMARY:
Clinical Retina research studies often collect aqueous samples in hopes of estimating levels of drug or cytokines in the vitreous. Little is known about how well vitreous and aqueous correlate. This study will collect vitreous and aqueous samples at the same time to evaluate and compare drug and cytokine levels.

The overall objective of this study is to evaluate the molecular concentration of growth factors, cytokines and chemokines in human aqueous humor and vitreous samples collected from individuals undergoing pars plana vitrectomy for tractional retinal detachment secondary to proliferative diabetic retinopathy, exudative or tractional retinal detachment secondary to macular degeneration, macular hole or neovascular glaucoma.

DETAILED DESCRIPTION:
This is an open-label, pilot study of intravitreally administered ranibizumab in subjects undergoing pars plana vitrectomy (PPV) to repair tractional retinal detachment secondary to proliferative diabetic retinopathy, exudative serous retinal detachment, macular hole or neovascular glaucoma.

Consented, enrolled subjects will be eligible to receive a single open-label intravitreal injection of 0.5 mg ranibizumab administered prior to undergoing PPV if in the Retinal Specialists opinion there could be a benefit to the disease or procedure from ranibizumab therapy.

The proposed study will analyze aqueous humor and vitreous samples drawn at the same time during vitrectomy to evaluate the levels of growth factors, cytokines and chemokines from patients undergoing planned pars plana vitrectomy as part of their retinal care. For patients receiving ranibizumab, serum samples will also be collected to assess PK. Patients will be split into three groups based on diagnosis: Group 1: (ranibizumab) proliferative diabetic retinopathy (tractional retinal detachment), macular degeneration with exudative or tractional retinal detachment, macular hole or neovascular glaucoma. Group 1 may receive one injection of intravitreal ranibizumab 0.5mg prior to vitrectomy. The injection will be administered at least 1-14 days prior to vitrectomy. Group 2 will serve as the control group and will not receive intravitreal ranibizumab prior to surgery.

Aqueous humor, vitreous and serum samples will be obtained to measure and compare growth factor, cytokine, chemokine levels and ranibizumab levels (if received). Undiluted core vitreous biopsies will be taken at the start of victrectomy. Aproximately 1 mL of undiluted vitreous fluid will be obtained with a closed infusion line and by manual aspiration with cutting on through the vitrectomy probe into a 2.5 mL syringe connected along the aspiration line. The sample will be frozen immediately and stored at -80°C.

Approximately 100 microliters of aqueous humor will be collected prior to the start of vitrectomy through anterior chamber paracentesis in the peripheral clear cornea using a 27 gauge needle on a tuberculin microsyringe from the central papillary area. Aqueous is transferred to a vial and placed in liquid nitrogen upon removal from the anterior chamber. Aqueous humor samples are immediately frozen at -80°C within 2 hours of collection until transferred to outside laboratories for further analysis.

Serum samples will be obtained from patients in Group 1 at baseline (Day 0) prior to treatment with intravitreal ranibizumab and on the day of surgery prior to the start of vitrectomy. Serum samples will be processed according to Genentech standard operating procedures and samples will be frozen immediately at -80C until analysis is ready to begin.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Subjects with a diagnosis of tractional retinal detachment secondary to proliferative diabetic retinopathy, age-related macular degeneration with tractional or exudative retinal detachment, macular hole, epiretinal membrane, or neovascular glaucoma.

Exclusion Criteria:

* Subjects with history of vitrectomy in the study eye
* Presence of vitreous hemorrhage
* Subjects with history of laser photocoagulation in the study eye within 3 months of vitrectomy
* Subjects unwilling to undergo pars plana vitrectomy
* Subjects unwilling to receive intravitreal ranibizumab prior to pars plana vitrectomy unless diagnosis of macular hole or epiretinal membrane
* Subjects who may need or have received systemic anti-VEGF for oncology in the past year
* Subjects with history of anti-VEGF injection within 4 months before vitrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Cytokine Levels | Collected at Baseline
  Growth factor, cytokine, chemokine , and ranibizumab (if applicable) concentration in aqueous and vitreous samples collected during pars plana vitrectomy

SECONDARY OUTCOMES:
Serum Pharmacokinetics | Up to Day 14
  Serum pharmacokinetic levels following a single intravitreal ranibizumab injection.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Avery, MD, Principal Investigator — California Retina Consultants
Locations (1):
- California Retina Consultants - Santa Barbara Office, Santa Barbara, California, United States